CLINICAL TRIAL: NCT03283566
Title: Hydroxychloroquine and Metabolic Outcomes in Patients Undergoing Total Pancreatectomy and Autologous Islet Transplantation: A Clinical, Molecular, and Genomic Study
Brief Title: Hydroxychloroquine and Metabolic Outcomes in Patients Undergoing TPAIT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute) (Other); Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 17-912
Record Dates: First submitted 2017-09-13; First posted 2017-09-14 (Actual); Results first posted 2022-03-11 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-04

CONDITIONS: Chronic Pancreatitis; Insulin Dependent Diabetes
Keywords: Pancreatectomy; Autologous Islet Transplantation; Pancreatitis; Diabetes; Hydroxychloroquine
MeSH Terms: conditions — Pancreatitis, Chronic; Diabetes Mellitus, Type 1; Pancreatitis; Diabetes Mellitus | interventions — Hydroxychloroquine

STUDY DESIGN:
Intervention Model Description: open label, randomized, two-arm, single-blinded, placebo-controlled, parallel
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The study will be single-blinded. The PI, biostatistician who will analyze the data, consultants, and technicians running assays will be blinded to the study arm into which the subjects have been randomized. An alphanumeric identifier that refers to the study subject without any indicators of study arm allocation will be used. Only the surgeons and the research coordinator, but not the personnel conducting the metabolic studies, will be un-blinded as to the study arm randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hydroxychloroquine (Active Comparator): Administered pre-transplant through 3 months after surgery.
  Interventions: Drug: Hydroxychloroquine
- Placebo (Placebo Comparator): Placebo treatment following the same schedule as Arm 1 (i.e. Hydroxychloroquine).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hydroxychloroquine — Subjects will receive a pre-transplant 200 mg daily dose of HCQ 30 days before TPAIT and will continue on the drug for 3 months after surgery.
  Other Names: Plaquenil
  Arms: Hydroxychloroquine
Drug: Placebo — Subjects will receive a pre-transplant placebo 30 days before TPAIT and will continue on the placebo for 3 months after surgery.
  Arms: Placebo

SUMMARY:
This will be a pilot, 12-month phase II, open label, randomized, two-arm, single-blinded, placebo-controlled, parallel clinical trial of individuals undergoing TPAIT (Total Pancreatectomy and Autologous Islet Transplantation) for treatment of chronic pancreatitis (CP). The two study arms consist of HCQ-treated (Hydroxychloroquine) and placebo-treated individuals. The purpose of this study is to investigate the effects of HCQ administration compared to placebo on islet cell function post-autologous transplantation.

DETAILED DESCRIPTION:
A compelling level of evidence exists on the effects of the innate immunity-driven inflammation on the decline of functional beta cell mass in the autologous transplant setting. The investigators hypothesize that HCQ administration during the peri-transplant period will preserve islet mass and improve islet cell function in TPAIT by reducing inflammation. The investigators specifically aim to demonstrate a higher stimulated C-peptide level as well as greater glucose control in response to mixed meal tolerance testing (MMTT) at 6 and 12 months following TPAIT in patients treated with HCQ compared to placebo. A better response in the HCQ arm suggests improved islet survival and metabolic performance, potentially facilitating higher rates of insulin independence.

HCQ administration:

Arm 1 (n=5): Subjects will receive a pre-transplant HCQ 200 mg daily dose 30 days prior TPAIT followed by HCQ use for an additional 3 months post-surgery.

Arm 2 (n=5) subjects will receive placebo treatment following the same schedule as in Arm 1.

Exploratory mechanistic studies:

All subjects will undergo a MMTT to assess islet cell function at 6 and 12 months following TPAIT (in addition to MMTT pre-surgery performed as standard of care, and whose results will be used for pre-randomization in this pilot). Baseline metabolic tests obtained too early after surgery may not be indicative of islet function, due to insulin supporting therapy administered for several weeks after transplantation. Also, compelling data indicate that stabilization of islet function may require up to 1 year to occur. Blood glucose and C-peptide serum levels will be measured in peripheral blood samples immediately prior and subsequent to MMTT. The research coordinator will contact the subjects at 3, 6 and 12 months for interview on the course of follow up and will assist in scheduling the 6 and 12-month appointments for MMTT.

Mitochondrial Function and Metabolic Outcomes in TPAIT:

Mitochondrial efficiency is important in the setting of TPAIT, where increase in metabolic demand and decrease in oxygenation have been established. The investigators will assess mitochondrial efficiency by measuring rates of mitochondrial respiration and glycolysis. These measures will be obtained on islets procured for donation and after islet isolation. Small amounts of digest left after islet isolation, that would normally be discarded, will be used for this portion of the study. The islets from the digest will be collected and will undergo extracellular efflux analysis through the Seahorse XF analyzer for mitochondrial function assessment. Commercially available normal human islet cells for experiments will be used as control. Controls will be compared simultaneously with islets isolated from study subjects.

Genome-wide Gene Expression in TPAIT Patients:

On the genomic level, several genetic pathways have been implicated in islet cell function and survival. The genetic profiles of islet cells from CP patients undergoing TPAIT have not been evaluated yet. The investigators aim to build an RNA-gene sequence database for islet cells of CP patients undergoing TPAIT, specifically targeting genes previously identified as key players in islet function. Small amounts of digest from the procedure used for isolating islets, and what remains in the circuit after the isolation process is complete, that would normally be discarded, will also be used for islet gene expression assessment.

ELIGIBILITY:
Inclusion Criteria:

* Clinically confirmed diagnosis of chronic pancreatitis (CP)
* Intractable abdominal pain
* History of failed operation(s) for CP
* Recurrent acute pancreatitis
* HbA1c <8.0%
* Sustained alcohol remission
* Chronic narcotic use

Exclusion Criteria:

* Insulin dependence
* Pancreatic carcinoma
* Pancreatic mass suspicious for carcinoma
* Cirrhosis
* Portal hypertension
* Continued alcohol abuse
* Manufacturer's product label-contraindicated use of HCQ
* History of retinopathy
* Actual weight at enrollment <40 Kg

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-10-03 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Betul Hatipoglu, MD, Principal Investigator — Staff
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hydroxychloroquine | Placebo
Started | 4 | 5
Completed | 3 | 3
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hydroxychloroquine | Placebo | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 6
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (12) | 37 (3) | 43.5 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 0 | 2 | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Quotient of Stimulated C-peptide/Glucose Level Normalized for IEQ/Kg Infused in Response to MMTT
Description: HCQ-treated compared to placebo arm. This outcome measure was reported in Mean and Standard deviation looking at C peptide/glucose secretion at 90 mins during mixed meal test adjusted for IEG/Kg (islet cell equivalency) infused to the patient.
Time Frame: 12 months
Population: C-peptide/Glucose = ng/mg glucose/IEQ/kg - Primary 12-month endpoint
Measure: Mean (Standard Deviation); unit: ng/mg glucose/IEQ/kg
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 3 | 3
ng/mg glucose/IEQ/kg | .000000077 (.000000096) | 0.000000079 (.00000012)

2. Secondary Outcome: C-peptide AUC Response to MMTT
Description: HCQ-treated compared to placebo arm. We used a standard, 5 hour Mixed meal tolerance test (MMT). Blood draws were taken every 15 mins for the first hours, then every 30 mins the second hour, then hourly until completion.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: ng/mL/min
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 3 | 3
ng/mL/min | 813 (463) | 588 (391)
Statistical Analysis 1: Comparison: Hydroxychloroquine vs Placebo; Test type: Equivalence — Assuming a 20-30% difference in outcome (CP/G quotient) between study arms, which is equivalent to 0.08-0.12 CP/G difference and a 0.07 standard deviation, a sample size of 6 subjects (1:1 randomization) will detect a CP/G difference of at least 0.12, assuming 80% power, with a 0.05 significance level; p = 0.739, ANOVA

3. Secondary Outcome: Ratio of C-peptide AUC to Glucose AUC in Response to MMTT Adjusted for Infused Islet Cell Mass
Description: C-peptide, ng/mL/min/IEQ/kg iAUC post-MMTT. Our measurement can be reported in area under the curve for C-peptide normalized for glucose values as well as Islet cell mass infused to the patient in order to compare placebo vs intervention arms.
Time Frame: 12 months
Population: Treatment versus placebo
Measure: Mean (Standard Deviation); unit: ng/mL/min/IEQ/kg iAUC post-MMT
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 3 | 3
ng/mL/min/IEQ/kg iAUC post-MMT | 0.00091 (0.0006) | 0.00222 (0.0029)

ADVERSE EVENTS:
Time Frame: About 3 years total study time. Each patient was assessed during a period of 12 months.
Description: No difference from clinicaltrials.gov definitions
Arm/Group | Hydroxychloroquine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 0/3 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-25): https://cdn.clinicaltrials.gov/large-docs/66/NCT03283566/Prot_SAP_000.pdf